CLINICAL TRIAL: NCT01574690
Title: Correlation of Physical Exam Versus Non-invasive Near-infrared Spectroscopy Versus Invasive Hemodynamic Assessment of Central Venous Pressure
Brief Title: Correlation of Physical Exam Versus Non-invasive Assessment Versus Invasive Assessment of Central Venous Pressure
Status: Completed | Type: Observational
Sponsor: Mespere Lifesciences Inc. (Industry)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Other Study IDs: MLS STP-9000008; HUM00054670 (Other: University of Michigan)
Record Dates: First submitted 2012-04-05; First posted 2012-04-10 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Central Venous Pressure
Keywords: central venous pressure; right heart catheter (RHC); non-invasive monitor; physical exam of jugular venous pressure; heart failure (HF)
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart failure patients: 50 subjects (both male and female) Heart failure patients already receiving RHC as part of their usual care
  Interventions: Device: Mespere Venus System; Procedure: Right heart catheterization (RHC); Procedure: Physical examination of jugular vein

INTERVENTIONS:
Device: Mespere Venus System — For this non-invasive system, an adhesive patch (connected to the Mespere Venus system) is placed on the neck of the subject, to determine if the CVP values displayed by the device correlates with the CVP values obtained by RHC and physical exam
  Other Names: Non-invasive central venous pressure system
Procedure: Right heart catheterization (RHC) — Invasive procedure to assess CVP. Standard of care.
Procedure: Physical examination of jugular vein — Physicians assess CVP using the subject's jugular vein.
  Other Names: Jugular venous pressure (JVP)

SUMMARY:
The purpose of this study is to establish the accuracy of a non-invasive device that uses near infrared spectroscopy (NIRS) to estimate central venous pressure (CVP) comparing it to physical exam and invasive hemodynamic measurement via right heart catheterization (RHC).

DETAILED DESCRIPTION:
Estimation of volume status is crucial when making treatment decisions for heart failure patients. Volume status is often assessed clinically by estimating the CVP, which is an estimate of right atrial filling pressure, by assessing the level of jugular venous distention. This method is quick and non-invasive but can be prone erroneous measurement due to human error and limitations secondary to body habitus and anatomical variation.

RHC is a procedure used for invasive hemodynamic measurement commonly used in heart failure patients. CVP can be measured directly via RHC using a pulmonary artery catheter. It is considered the gold standard for measuring intra-cardiac filling pressures and calculation of cardiac output and pulmonary and systemic vascular resistance. The obvious downside of RHC is that is invasive, time consuming, and has many potential serious risks including vascular complication, pneumothorax, infection, arrhythmia, valvular damage, etc.

A non-invasive, quick, and accurate way to estimate central venous pressure and oximetry could benefit patient care. NIRS is an optical imaging technology that has been proposed to estimate central venous pressure non-invasively. Our intent is to determine the accuracy of NIRS in assessment of CVP using the Mespere Venus device.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Heart failure patients already receiving RHC as part of their usual care
* Signed written and informed consent

Exclusion Criteria:

* Lack of patient consent
* Presence of known anatomical shunt or AV dialysis fistula
* Sepsis, fever
* Anemia (Hgb < 10)
* Allergy to adhesive tape
* Known central vein stenosis
* Previous cardiac transplant
* Unable to identify external jugular vein
* Ongoing photodynamic therapy
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with heart failure (HF)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Central Venous Pressure (CVP) | 0-3 hours
  To determine if the CVP from the non-invasive monitor correlates with the CVP from the invasive method (via RHC) and/or the CVP from the physical exam

CONTACTS AND LOCATIONS:
Overall Officials: Todd M Koelling, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Cardiovascular Center, Ann Arbor, Michigan, United States